CLINICAL TRIAL: NCT01590277
Title: Ability of Partial Inverse Agonist, Iomazenil, to Block Ethanol Effects in Humans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CLIN-026-11F
Record Dates: First submitted 2012-04-30; First posted 2012-05-02 (Estimated); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-09

CONDITIONS: Active Ethanol and Active Iomazenil; Active Ethanol and Placebo Iomazenil; Placebo Ethanol and Active Iomazenil; Placebo Ethanol and Placebo Iomazenil; Alcohol Effect; Driving Under the Influence; Alcohol Impairment
MeSH Terms: conditions — Driving Under the Influence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Active Ethanol and Active Iomazenil (Experimental): Participants will receive in a randomized, double-blind, cross-over design, ethanol or placebo and iomazenil or placebo.
  Potential Randomizations: a) active ethanol and placebo iomazenil, b) active ethanol and active iomazenil, c) placebo ethanol and active iomazenil, and d) placebo ethanol and placebo iomazenil
  Interventions: Drug: Active Ethanol; Drug: Active Iomazenil
- Active Ethanol and Placebo Iomazenil (Experimental): Participants will receive in a randomized, double-blind, cross-over design, ethanol or placebo and iomazenil or placebo.
  Potential Randomizations: a) active ethanol and placebo iomazenil, b) active ethanol and active iomazenil, c) placebo ethanol and active iomazenil, and d) placebo ethanol and placebo iomazenil
  Interventions: Drug: Active Ethanol; Drug: Placebo
- Placebo Ethanol and Active Iomazenil (Experimental): Participants will receive in a randomized, double-blind, cross-over design, ethanol or placebo and iomazenil or placebo.
  Potential Randomizations: a) active ethanol and placebo iomazenil, b) active ethanol and active iomazenil, c) placebo ethanol and active iomazenil, and d) placebo ethanol and placebo iomazenil
  Interventions: Drug: Active Iomazenil; Drug: Placebo
- Placebo Ethanol and Placebo Iomazenil (Placebo Comparator): Participants will receive in a randomized, double-blind, cross-over design, ethanol or placebo and iomazenil or placebo.
  Potential Randomizations: a) active ethanol and placebo iomazenil, b) active ethanol and active iomazenil, c) placebo ethanol and active iomazenil, and d) placebo ethanol and placebo iomazenil
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Active Ethanol — Target BrAC of 0.1% reached over 30 minutes and then clamped to maintain this dose for an additional 60 minutes. This dose is equivalent to consuming approximately 5 drinks. Administered over a total of 90 minutes.
  Arms: Active Ethanol and Active Iomazenil; Active Ethanol and Placebo Iomazenil
Drug: Active Iomazenil — Active iomazenil, administered intravenously at a dose of 3.7 ug/kg. Administered over 10 minutes, beginning 10 minutes after the start of the ethanol/placebo clamp.
  Arms: Active Ethanol and Active Iomazenil; Placebo Ethanol and Active Iomazenil
Drug: Placebo — Control: no alcohol, administered for a total of 90 minutes.
  Arms: Placebo Ethanol and Active Iomazenil; Placebo Ethanol and Placebo Iomazenil
Drug: Placebo — Control: no iomazenil, administered for a total of 10 minutes
  Arms: Active Ethanol and Placebo Iomazenil; Placebo Ethanol and Placebo Iomazenil

SUMMARY:
Alcohol is abused commonly, but there is no remedy for alcohol intoxication. This project is looking at the substance iomazenil and its effect on alcohol intoxication and alcohol's effects on driving using a driving simulator.

DETAILED DESCRIPTION:
Alcohol is abused commonly, but there is no antidote for alcohol intoxication the way naltrexone or naloxone is an antidote for opioids. A medication that has the potential to block alcohol actions in the Central Nervous System could act as a unique medication in the treatment of alcohol intoxication and alcoholism. This project is evaluating the benzodiazepine partial inverse agonist, iomazenil, as an agent that could reverse alcohol's effects on subjective intoxication, alcohol's effects on driving using a driving simulator and on measures of electrophysiology in the laboratory in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Males
* 21-35 years old
* Medically healthy

Exclusion Criteria:

* Under the age of 21 or greater than the age 35
* History of seizures

Ages: 21 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2012-12-14 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2018-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deepak C D'Souza, MD MBBS, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (1):
- VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 33 participants initiated study procedures beyond screening. Of these 33 participants, 30 completed all four test days (thus receiving all four treatment conditions, one on each of the four test days), 2 participants withdrew from the study after 2 test days (receiving 2 out of the 4 treatment conditions), and 1 participant withdrew after 1 test day (receiving 1 out of the 4 treatment conditions..
Pre-assignment Details: Each participant will receive in a randomized, double-blind, cross-over design, ethanol or placebo and iomazenil or placebo.
  Potential randomizations for each test day: a) active ethanol and placebo iomazenil, b) active ethanol and active iomazenil, c) placebo ethanol and active iomazenil, and d) placebo ethanol and placebo iomazenil
Groups:
- All Study Participants: ARM 1: Active Ethanol and Active Iomazenil:
  Active Ethanol: Target BrAC of 0.1% reached over 30 minutes and then clamped to maintain this dose for an additional 60 minutes. This dose is equivalent to consuming approximately 5 drinks. Administered over a total of 90 minutes.
  Active Iomazenil: Active iomazenil, administered intravenously at a dose of 3.7 ug/kg. Administered over 10 minutes, beginning 10 minutes after the start of the ethanol/placebo clamp.
  ARM 2: Active Ethanol and Placebo Iomazenil
  Active Ethanol: Target BrAC of 0.1% reached over 30 minutes and then clamped to maintain this dose for an additional 60 minutes. This dose is equivalent to consuming approximately 5 drinks. Administered over a total of 90 minutes.
  Placebo: Control: no iomazenil, administered for a total of 10 minutes
  ARM 3: Placebo Ethanol and Active Iomazenil.
  Active Iomazenil: Active iomazenil, administered intravenously at a dose of 3.7 ug/kg. Administered over 10 minutes, beginning 10 minutes after the start of the ethanol/placebo clamp.
  Placebo: Control: no alcohol, administered for a total of 90 minutes.
  ARM 4: Placebo Ethanol and Placebo Iomazenil
  Placebo: Control: no alcohol, administered for a total of 90 minutes.
  Placebo: Control: no iomazenil, administered for a total of 10 minutes
Period: Overall Study
Arm/Group | All Study Participants
Started | 33
Active Ethanol and Placebo Iomazenil | 31
Active Ethanol and Active Iomazenil | 30
Placebo Ethanol and Active Iomazenil | 32
Placebo Ethanol and Placebo Iomazenil | 32
Completed | 26
Not Completed | 7
Not completed — Withdrawal by Subject | 3
Not completed — Withdrawal by Subject | 2
Not completed — Withdrawal by Subject | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Enrolled Participants (N=33): Baseline demographics for all participants that initiated study procedures beyond screening.
  Participants will receive in a randomized, double-blind, cross-over design, ethanol or placebo and iomazenil or placebo on each of 4 separate test days. Potential Randomizations for each test day are: a) active ethanol and placebo iomazenil, b) active ethanol and active iomazenil, c) placebo ethanol and active iomazenil, and d) placebo ethanol and placebo iomazenil. A participant who completes all four test days will receive each of the potential randomizations throughout their study participation.
Arm/Group | Enrolled Participants (N=33)
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 33
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.76 (3.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 26
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Biphasic Ethanol Effects Scale (BAES)
Description: A 14-item scale with 7 items designated to assess stimulant effects associated with the ascending limb of ethanol intoxication and 7 items developed to measure sedative effects associated with the descending limb of ethanol intoxication. The BAES full scale would be 0 to 140. However, the scale itself is analyzed by breaking up the full 14 item scale into 2 parts - sedation and stimulation. Therefore, the total score for sedation ranges from 0 to 70, with higher scores indicating more sedation, and the total score for stimulation also ranges from 0 to 70, with higher scores indicating more stimulation.
  Timepoints: Administered 160 mins (M160) and 10 mins (M10) prior to the target ethanol/placebo dose being reached, when the target ethanol dose (BrAC of 0.1%)/placebo has been reached (0), and 15 (P15), 70 (P70), 90 (P90), and 150 (P150) minutes after the target ethanol/placebo dose has been reached.
Time Frame: Administered 160 mins and 10 mins prior to the target ethanol/placebo dose being reached, when the target ethanol dose (BrAC of 0.1%)/placebo has been reached, and 15, 70, 90, 150, and 240 minutes after the target ethanol/placebo dose has been reached.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Active Ethanol and Active Iomazenil: Each participant will receive in a randomized, double-blind, cross-over design, ethanol or placebo and iomazenil or placebo.
  Potential randomizations for each test day: a) active ethanol and placebo iomazenil, b) active ethanol and active iomazenil, c) placebo ethanol and active iomazenil, and d) placebo ethanol and placebo iomazenil
  Active Ethanol: Target BrAC of 0.1% reached over 30 minutes and then clamped to maintain this dose for an additional 60 minutes. This dose is equivalent to consuming approximately 5 drinks. Administered over a total of 90 minutes.
  Active Iomazenil: Active iomazenil, administered intravenously at a dose of 3.7 ug/kg. Administered over 10 minutes, beginning 10 minutes after the start of the ethanol/placebo clamp.
- Active Ethanol and Placebo Iomazenil: Each participant will receive in a randomized, double-blind, cross-over design, ethanol or placebo and iomazenil or placebo.
  Potential randomizations for each test day: a) active ethanol and placebo iomazenil, b) active ethanol and active iomazenil, c) placebo ethanol and active iomazenil, and d) placebo ethanol and placebo iomazenil
  Active Ethanol: Target BrAC of 0.1% reached over 30 minutes and then clamped to maintain this dose for an additional 60 minutes. This dose is equivalent to consuming approximately 5 drinks. Administered over a total of 90 minutes.
  Placebo: Control: no iomazenil, administered for a total of 10 minutes
- Placebo Ethanol and Active Iomazenil: Each participant will receive in a randomized, double-blind, cross-over design, ethanol or placebo and iomazenil or placebo.
  Potential randomizations for each test day: a) active ethanol and placebo iomazenil, b) active ethanol and active iomazenil, c) placebo ethanol and active iomazenil, and d) placebo ethanol and placebo iomazenil
  Active Iomazenil: Active iomazenil, administered intravenously at a dose of 3.7 ug/kg. Administered over 10 minutes, beginning 10 minutes after the start of the ethanol/placebo clamp.
  Placebo: Control: no alcohol, administered for a total of 90 minutes.
- Placebo Ethanol and Placebo Iomazenil: Each participant will receive in a randomized, double-blind, cross-over design, ethanol or placebo and iomazenil or placebo.
  Potential randomizations for each test day: a) active ethanol and placebo iomazenil, b) active ethanol and active iomazenil, c) placebo ethanol and active iomazenil, and d) placebo ethanol and placebo iomazenil
  Placebo: Control: no alcohol, administered for a total of 90 minutes.
  Placebo: Control: no iomazenil, administered for a total of 10 minutes
Arm/Group | Active Ethanol and Active Iomazenil | Active Ethanol and Placebo Iomazenil | Placebo Ethanol and Active Iomazenil | Placebo Ethanol and Placebo Iomazenil
Number analyzed (Participants) | 30 | 31 | 32 | 32
score on a scale
  Sedation Effects (Timepoint M160) | 3.767 (6.826) | 3.935 (7.771) | 3.813 (7.368) | 3.194 (5.431)
  Sedation Effects (Timepoint M10) | 4.767 (5.74) | 4.484 (6.623) | 3.438 (5.853) | 3.968 (7.092)
  Sedation Effects (Timepoint 0) | 5.267 (5.271) | 5.258 (6.153) | 2.875 (5.74) | 3.452 (6.35)
  Sedation Effects (Timepoint P15) | 7 (7.409) | 5.677 (7.368) | 6.75 (8.74) | 3.387 (6.249)
  Sedation Effects (Timepoint P70) | 7.2 (11.075) | 6.806 (9.393) | 3.469 (6.17) | 2.516 (5.092)
  Sedation Effects (Timepoint P90) | 4.9 (6.088) | 5.677 (8.89) | 2.875 (6.384) | 1.452 (3.491)
  Sedation Effects (Timepoint P150) | 2.586 (4.594) | 4.567 (7.257) | 2.813 (5.688) | 1.548 (3.897)
  Stimulation Effects (Timepoint M160) | 11.2 (11.152) | 13 (13.844) | 13.281 (12.606) | 12.387 (11.292)
  Stimulation Effects (Timepoint M10) | 12.567 (12.297) | 12.903 (11.47) | 12.188 (12.678) | 9.129 (9.57)
  Stimulation Effects (Timepoint 0) | 13.767 (12.813) | 14.484 (13.466) | 10.406 (12.018) | 8.065 (9.352)
  Stimulation Effects (Timepoint P15) | 12.8 (13.697) | 13.968 (12.875) | 9.625 (11.187) | 8.452 (9.305)
  Stimulation Effects (Timepoint P70) | 9.233 (11.193) | 9.839 (11.827) | 10.125 (11.853) | 9.903 (11.324)
  Stimulation Effects (Timepoint P90) | 8.833 (10.449) | 9.742 (12.762) | 10.094 (11.217) | 9.71 (11.261)
  Stimulation Effects (Timepoint P150) | 8.793 (11.004) | 9.867 (13.32) | 10.406 (11.67) | 9.484 (9.743)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected beginning at the time of screening and for each of the four test days, through to the completion of the study. Follow up data was obtained at 1 week, 1 month, 6 months, and 1 year following the last test day.
Description: Adverse events are reported for each test day condition.
Arm/Group | Active Ethanol and Active Iomazenil | Active Ethanol and Placebo Iomazenil | Placebo Ethanol and Active Iomazenil | Placebo Ethanol and Placebo Iomazenil
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/31 | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/31 | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 3/30 | 1/31 | 3/32 | 0/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Ethanol and Active Iomazenil (N=30) | Active Ethanol and Placebo Iomazenil (N=31) | Placebo Ethanol and Active Iomazenil (N=32) | Placebo Ethanol and Placebo Iomazenil (N=32)
Lightheaded (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Stomach Cramps (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-06-10): https://cdn.clinicaltrials.gov/large-docs/77/NCT01590277/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-10): https://cdn.clinicaltrials.gov/large-docs/77/NCT01590277/SAP_001.pdf